CLINICAL TRIAL: NCT01180803
Title: Efficacy of Oxygen Therapy Delivered by Systems Using Oxygen-Saving Valves in COPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche (Other)
Responsible Party: Principal Investigator, DELRIEU Jacqueline, Clinical Project Manager, Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EVAL- CLIN A00690-39
Record Dates: First submitted 2010-08-11; First posted 2010-08-12 (Estimated); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: LUNG DISEASES, OBSTRUCTIVE
Keywords: COPD - long term oxygenotherapy; COPD patients with respiratory failure
MeSH Terms: conditions — Lung Diseases, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- oxygen-saving valves (Experimental)
  Interventions: Device: pulse oxygen supplementation devices
- continuous oxygen supplementation (Active Comparator)
  Interventions: Device: continuous oxygen

INTERVENTIONS:
Device: pulse oxygen supplementation devices — oxygen therapy delivered by systems using oxygen-saving valves
  Other Names: pulse group
  Arms: oxygen-saving valves
Device: continuous oxygen — oxygen therapy delivered by continuous liquid oxygen devices
  Other Names: continuous group
  Arms: continuous oxygen supplementation

SUMMARY:
The purpose of this study is to compare the efficacy of oxygen therapy delivered by systems using oxygen-saving valves or not (continuous oxygen). We aim to determine if systems using oxygen-saving valves are equally effective as continuous oxygen delivery systems in reducing exercise-induced hypoxemia in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* COPD on necessity of long term oxygen therapy
* Able to give their written consent

Exclusion Criteria:

* Unstable patients with COPD
* Patients with restrictive respiratory disease
* Patients with cardiac or neurologic disease contre-indicating the different evaluations

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-07; Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
oxygen saturation during 6 minutes walking test | 1 day

SECONDARY OUTCOMES:
Walking distance during the 6 minutes walking test | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Fédération ANTADIR, Paris, France